CLINICAL TRIAL: NCT04868877
Title: Phase 1/2 Dose Escalation and Expansion Study Evaluating MCLA-129, a Human Anti-EGFR and Anti-c-MET Bispecific Antibody, in Patients With Advanced NSCLC and Other Solid Tumors
Brief Title: Phase 1/2 Study Evaluating MCLA-129, a Human Anti-EGFR, Anti-c-MET Bispecific Antibody, in Advanced NSCLC and Other Solid Tumors, Alone and in Combination
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-129-CL01
Record Dates: First submitted 2021-04-09; First posted 2021-05-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer Metastatic; Gastric Cancer; Esophageal Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma; Colorectal Cancer
Keywords: MCLA-129; EGFR inhibitor; NSCLC; C-MET; GC/GEJ; Head and Neck Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Head and Neck Neoplasms | interventions — osimertinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part 2 NSCLC Second-line or more harboring EGFR exon 20 Insertion (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks at the recommended Phase II dose (RP2D).
  Interventions: Drug: MCLA-129
- Part 2 NSCLC Second-line or more harboring cMet exon 14 skipping mutation (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks at the recommended Phase II dose (RP2D).
  Interventions: Drug: MCLA-129
- Part 2 Selected solid tumors with or without an EGFR or cMet alteration (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks at the recommended Phase II dose (RP2D).
  Interventions: Drug: MCLA-129
- Part 2 NSCLC First-line harboring EGFR sensitizing mutations (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks at the recommended Phase II dose (RP2D) and Osimertinib orally once daily starting at a dose of 80mg.
  Interventions: Drug: MCLA-129; Drug: Osimertinib
- Part 2 NSCLC Second-line or more, osimertinib resistant (combo with osimertinib) (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks at the recommended Phase II dose (RP2D) and Osimertinib orally once daily starting at a dose of 80mg.
  Interventions: Drug: MCLA-129; Drug: Osimertinib
- Part 2 NSCLC Second-line or more, osimertinib resistant (combo with chemotherapy) (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks at the recommended Phase II dose (RP2D) and chemotherapy every three weeks per standard of care according to local guidance.
  Interventions: Drug: MCLA-129; Drug: Chemotherapy
- Part 2 NSCLC Third-line or more, osimertinib resistant, platinum resistant (combo with chemotherapy) (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks at the recommended Phase II dose (RP2D) and chemotherapy every three weeks per standard of care according to local guidance.
  Interventions: Drug: MCLA-129; Drug: Chemotherapy

INTERVENTIONS:
Drug: MCLA-129 — full length IgG1 bispecific antibody that specifically targets the receptor tyrosine kinases EGFR and c-MET
  Other Names: bispecific
Drug: Osimertinib — Approved, 3rd-generation EGFR-TKI
  Other Names: Tagrisso
  Arms: Part 2 NSCLC First-line harboring EGFR sensitizing mutations; Part 2 NSCLC Second-line or more, osimertinib resistant (combo with osimertinib)
Drug: Chemotherapy — administrated by IV infusion
  Arms: Part 2 NSCLC Second-line or more, osimertinib resistant (combo with chemotherapy); Part 2 NSCLC Third-line or more, osimertinib resistant, platinum resistant (combo with chemotherapy)

SUMMARY:
A phase 1/2 open-label multicenter study will be performed with an initial dose escalation part to determine the MTD and/or the RP2D of MCLA-129 in monotherapy or in combination in patients with NSCLC, HNSCC, GC/GEJ, ESCC, or other solid tumors and who are treatment naïve or have progressed after receiving prior therapy for advanced/metastatic disease.

ELIGIBILITY:
Part One: Patients with NSCLC, GC/GEJ, HNSCC, or ESCC who have failed prior standard first-line treatment. Patients must have progressed on or be intolerant to therapies that are known to provide clinical benefit. There is no limit to the number of prior treatment regimens.

Part Two: Patients with NSCLC, HNSCC, other solid tumors and applicable mutations as determined by the investigator.

* Availability of archival or a fresh tumor tissue sample.
* Measurable disease as defined by RECIST version 1.1 by radiologic methods.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥ 12 weeks, as per Investigator.
* Adequate organ function (as per protocol)

Exclusion Criteria:

* Central nervous system metastases that are untreated or symptomatic, or require radiation, surgery, or continued steroid therapy (> 10 mg prednisone or equivalent) to control symptoms within 14 days of study entry.
* Known leptomeningeal involvement.
* Participation in another clinical study or treatment with any investigational drug within 4 weeks prior to study entry.
* Systemic anticancer therapy or immunotherapy within 4 weeks or 5 half-lives, whichever is shorter, of the first dose of study drug. For cytotoxic agents that have major delayed toxicity (e.g., mitomycin C, nitrosoureas), a washout period of 6 weeks is required.
* Major surgery or radiotherapy within 3 weeks of the first dose of study drug. Patients who received prior radiotherapy to ≥25% of bone marrow at any time are not eligible.
* Persistent grade >1 clinically significant toxicities related to prior antineoplastic therapies (except for alopecia); stable sensory neuropathy ≤ grade 2 NCI-CTCAE v5.0 and hypothyroidism ≤ grade 2 which is stable on hormone replacement are allowed.
* History of hypersensitivity reaction or any toxicity attributed to human proteins or any of the excipients that warranted permanent cessation of these agents. History of hypersensitivity reaction or any toxicity attributed to chemotherapy and components.
* History of clinically significant cardiovascular disease
* Past medical history of ILD or pneumonitis, or any evidence of clinically active ILD or pneumonitis.
* Previous or concurrent malignancy, excluding non-basal cell carcinomas of skin or carcinoma in situ of the uterine cervix, unless the tumor was treated with curative or palliative intent and in the opinion of the Investigator, with Sponsor agreement, the previous or concurrent malignancy condition does not affect the assessment of safety and efficacy of the study drug.
* Current serious illness or medical conditions including, but not limited to uncontrolled active infection, clinically significant pulmonary, metabolic or psychiatric disorders
* Active Hepatitis B infection without receiving antiviral treatment.
* Positive test for Hepatitis C
* Known history of HIV (HIV 1/2 antibodies). Patients with HIV with undetectable viral load are allowed. In

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) | First 28 days of treatment
  To determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of single-agent MCLA-129 as well as in combination with chemotherapy in patients with NSCLC, GC/GEJ adenocarcinoma, HNSCC or ESCC, with disease progression after prior therapy for advanced/metastatic disease.
To evaluate clinical activity, as assessed by ORR | From first dose until RECIST progression or initiation of an alternative treatment, whichever occurs first.
  To evaluate the ORR of MCLA-129 monotherapy or in combination with an EGFR TKI or chemotherapy in molecularly defined populations of advanced/metastatic solid tumors.

SECONDARY OUTCOMES:
To evaluate preliminary antitumor activity in terms of BOR | From first dose until RECIST progression or initiation of an alternative treatment, whichever occurs first.
  To evaluate preliminary antitumor activity of MCLA-129 monotherapy as well as in combination with an EGFR TKI or chemotherapy in terms of best overall response (BOR)
To evaluate preliminary antitumor activity in terms of DCR | From first dose until RECIST progression or initiation of an alternative treatment, whichever occurs first.
  To evaluate preliminary antitumor activity of single-agent MCLA-129 as well as in combination with an EGFR TKI or with chemotherapy in terms of Disease Control Rate (DCR).
To evaluate preliminary antitumor activity in terms of DoR | From first dose until RECIST progression or initiation of an alternative treatment, whichever occurs first.
  To evaluate preliminary antitumor activity of single-agent MCLA-129 as well as in combination with an EGFR TKI or with chemotherapy in terms of Duration of Response (DoR)
To evaluate progression-free survival (PFS) | From first dose until RECIST progression or until 1 year after treatment, whichever occurs first.
  To evaluate progression-free survival (PFS) of single-agent MCLA-129 as well as in combination with an EGFR TKI or with chemotherapy.
To evaluate overall survival (OS) | From first dose until RECIST progression or until 1 year after treatment, whichever occurs first.
  To evaluate overall survival (OS) of single-agent MCLA-129 as well as in combination with an EGFR TKI or with chemotherapy.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 of single-agent MCLA-129 as well as in combination with an EGFR TKI or with chemotherapy | From first dose until study treatment discontinuation
Proportion of patient with treatment discontinuations of single-agent MCLA-129 as well as in combination with an EGFR TKI or with chemotherapy. | From first dose until study treatment discontinuation
AE, regardless of relationship to study treatment | From first dose until study treatment discontinuation
All safety endpoints | From first dose until study treatment discontinuation
  including vital sign, lab, ECG, ECHO, 4 weeks CT scan, Eye exam

CONTACTS AND LOCATIONS:
Locations (51):
- United States (4):
  - University of California, Irvine, Orange, California
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - START Mountain Region, West Valley City, Utah
  - Next Oncology Virginia, Fairfax, Virginia
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - Antwerp University Hospital, Edegem
- France (12):
  - Clinique de l'Europe, Amiens
  - CHU Hopitaux de Bordeaux - Hôpital Saint-André, Bordeaux
  - CHU de Lyon - Louis Pradel Hospital, Bron
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Albert Calmette, Lille
  - L'Institut Paoli - Calmettes, Marseille
  - CHU de Nantes - Hôpital Nord Laennec, Nantes
  - Marie Wislez, Paris
  - Hôpital Bichat - Claude-Bernard, Paris
  - Hôpital Européen Georges Pompidou (HEGP), Paris
  - CHU de Poitiers, Poitiers
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
- Germany (2):
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - Sana Klinikum Offenbach GmbH, Offenbach
- Italy (8):
  - Istituto Nazionale dei Tumori Regina Elena, Roma, Rome
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - ASST degli Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Universitaria San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Netherlands (3):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- National Cancer Centre of Singapore, Singapore, Singapore
- South Korea (6):
  - Gachon University Gil Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei Cancer Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
- Spain (13):
  - Hospital HM Delfos, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - IOB Institute of Oncology - Hospital Quironsalud Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clínica Universidad de Navarra -Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Quirón Madrid, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Fundación Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No